CLINICAL TRIAL: NCT06147895
Title: A Randomized, Open-labelled, Parallel, Phase 1 Clinical Study to Evaluate the Safety, Reactogenicity and Immunogenicity of the Hepatitis B Vaccine CVI-HBV-002 in Adults
Brief Title: A Study to Evaluate the Safety, Reactogenicity and Immunogenicity of Prophylactic Hepatitis B Vaccine
Acronym: CVI-HBV-002
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CHA Vaccine Institute Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CVI-HBV-002-CT2001
Record Dates: First submitted 2023-11-15; First posted 2023-11-28 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2023-11

CONDITIONS: Vaccine-Preventable Diseases; Hepatitis B
MeSH Terms: conditions — Vaccine-Preventable Diseases; Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): CVI-HBV-002 1 mL Intramuscular injection at Baseline, Week 4, Week 8 / total 3 doses
  Interventions: Biological: CVI-HBV-002
- Group 2 (Experimental): CVI-HBV-002 1 mL Intramuscular injection at Baseline, Week 4, Week 24 / total 3 doses
  Interventions: Biological: CVI-HBV-002

INTERVENTIONS:
Biological: CVI-HBV-002 — Investigational Product

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of the investigational medicinal product, CVI-HBV-002.

DETAILED DESCRIPTION:
A Randomized, Open-labelled, Parallel, Phase 1 clinical study to evaluate the safety, reactogenicity and immunogenicity of the hepatitis B vaccine CVI-HBV-002 in adults

ELIGIBILITY:
Inclusion Criteria:

1. Any gender, age 19-64 years
2. Those whose anti-HBs titer is less than 10 mIU/mL
3. Those who have voluntarily agreed to participate in this clinical trial and signed the subject consent form

Exclusion Criteria:

1. Patient with positive test for antibody to hepatitis B core antigen (anti-HBc)
2. Acute illness and/or fever (tympanic temperature rises greater than 38 degrees Celsius) within 72 hours before administration of investigational product
3. A person who suffered from serious acute or chronic infection within 7 days prior to administration of investigational product (Those who need systemic antibiotic treatment or antiviral therapy)
4. In case of immunodeficiency or immune dysfunction, or if there is a family history of such
5. Patients with abnormal liver function test results
6. Patients with active bacterial, viral or fungal infections requiring systemic treatment
7. Patients with a history of serious heart disease (NYHA Functional Class III or IV heart failure, myocardial infarction within 6 months, ventricular tachyarrhythmias requiring treatment, or unstable angina, etc.)
8. Seizure disorders requiring anticonvulsant treatment
9. Patients with severe chronic obstructive pulmonary disease accompanied by hypoxemia
10. Patients with uncontrolled diabetes
11. Patients with uncontrolled hypertension
12. Patient with positive test for HBsAg, HIV or Hepatitis C
13. Those with hypersensitivity or anaphylactic reaction to HBV vaccine components
14. Those who have received immunosuppressive or immunomodulatory drugs within 6 months before screening
15. Patients who have received high-dose (20 mg or more per day based on prednisolone*) systemic corticosteroids for a long period of time (administration for more than 14 consecutive days) within 3 months before screening (in the case of topical corticosteroids, subject to the investigator's judgment)

    * Equivalent to cortisone 125 mg, hydrocortisone 100 mg, prednisone 20 mg, methylprednisolone 16 mg, triamcinolone 16 mg, dexamethasone 3 mg, betamethasone 2.4 mg
16. Patients currently undergoing hemodialysis
17. In case of continuous drinking (more than 21 units/week, 1 unit (1 cup) = 10g of pure alcohol) or alcohol dependence
18. In addition to the above, those who have clinically significant findings that are considered inappropriate for this study based on medical judgment by the principal investigator or person in charge
19. Pregnant or lactating women or self- and partner contraception during clinical trials (e.g., sterilization, intrauterine contraceptives, oral contraceptives in combination with interstitial barrier contraception, other hormone delivery systems in combination with interstitial barrier contraception, contraceptive cream, jelly or foam) Persons who cannot agree on diaphragms or condoms)
20. Patients who are concerned about the decline in daily function due to mental illness or who cannot understand the purpose and method of this clinical trial
21. Those who may show other serious febrile or systemic reactions
22. Those who are scheduled to participate in other clinical trials after being enrolled in this clinical trial, or who have participated in other clinical trials within 3 months before being enrolled in this clinical trial
23. Those who are considered difficult to conduct this clinical trial when judged by other investigators

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
Immediate adverse events | within 30 minutes post vaccination timepoint
  Occurrence of immediate adverse events
Solicited local and systemic signs and symptoms | Time Frame: Day 0 - Day 6 post each vaccination timepoint
  Occurrence, severity, and duration of solicited local injection site reactions for 7 days (Day 0-Day 6) following each vaccination. (e.g., pain in daily activities, redness and swelling in size(cm))
  Occurrence, severity, and duration of solicited systemic reactions for 7 days (Day 0-Day 6) following each vaccination. (e.g., myalgia, fatigue and headache in daily activities, fever in oral temperature)
Unsolicited signs and symptoms | Day 0-Day 28 post each vaccination timepoint
  Occurrence, severity, and relationship to vaccination of unsolicited adverse events until 28 days following each vaccination
SAEs | Up to Week 48 post the 3rd vaccination
  Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity
Safety as measured by clinical laboratory test, vial sign and physical examination parameters | Until Week 48 post the 3rd vaccination
  Occurrence, intensity, and relationship to vaccination of clinically significant adverse events

SECONDARY OUTCOMES:
Seroprotective Immune Response | Baseline, Weeks 4, 8, 12 and 56 for Group 1, baseline, Weeks 4, 8, 28 and 72 for Group 2
  Percentage of Subjects Who Have a Seroprotective Immune Response (Anti-HBsAg ≥ 10 Milli-international Unit (mIU)/mL) at baseline and at Weeks 4 post each vaccination and at last visit
Measurement of Serum GMT | Weeks 4, 8, 12 and 56 for Group 1, Weeks 4, 8, 28 and 72 for Group 2
  Serum GMT of Anti-HBsAg Measured at baseline and at Weeks 4 post each vaccination and at last visit

CONTACTS AND LOCATIONS:
Overall Officials: Youngsang Kim, Principal Investigator — CHA University Bundang Medical Center
Locations (1):
- CHA University Bundang Medical Center, Seongnam-si, Gyeonggi-do, South Korea